CLINICAL TRIAL: NCT04010734
Title: Primary Peroral Cholangioscopy Versus Endoscopic Retrograde Cholangiopancreatography (With Conventional Sampling - Brushing and Forceps Biopsy- Completed by Fluorescence In Situ Hybridization) in the Diagnosis of Biliary Strictures
Brief Title: Primary Cholangioscopy Versus ERCP in the Diagnosis of Biliary Strictures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Vincent Zoundjiekpon, principal investigator, University Hospital Olomouc
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: UHO001
Record Dates: First submitted 2019-06-01; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-06

CONDITIONS: Biliary Stricture
Keywords: suspected malignant biliary stricture; primary peroral cholangiscopy; endoscopic retrograde cholangiopancreatography; fluorescence in situ hybridization
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peroral Cholangioscopy examination (Active Comparator): Patient with suspected malignant biliary stricture (SMBS) is allowed:
  to the peroral Cholangioscopy examination with both visual and tissue diagnosis. The visual diagnosis is based on morphological and vascular patterns (presence or not of nodular or papilary masses, irregularity of the surface, morphology of the vessels and the fragility of mucosa). The tissue diagnosis consists on cytopathological evaluation after tissue sampling using minuature biopsy forceps (SpyBite). During this, 5-8 samples are taken under visual control, from different parts of the lesion.
  Interventions: Procedure: Peroral Cholangioscopy and Endoscopic retrograde cholangiopancreatography
- ERCP examination with sampling (Active Comparator): Patient with suspected malignant biliary stricture (SMBS) is allowed:
  to ERCP examination with both sampling by brushing and forceps biopsy, with subsequent pathological evaluation and an additional fluorescence in situ hybridization(FISH) examination of the specimens.
  ERCP (Endoscopic retrograde cholangiopancreatography) is the most widely used diagnostic procedure in patients with biliary obstruction. It enables to identify the biliary stricture, to determinate its location and help providing tissue sampling from the stricture for cytological evaluation. Brushing and endocanal forceps biopsies were the most used techniques, both with different specificity and sensitivity. It was demonstrated that Fluorescence in Situ Hybridization (FISH) improved the diagnostic yield of routine cytology. That is the reason why the investigators will combine FISH with the sampling methods to maximize the chance to make early diagnosis of the biliary stenosis.
  Interventions: Procedure: Peroral Cholangioscopy and Endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Procedure: Peroral Cholangioscopy and Endoscopic retrograde cholangiopancreatography — The peroral cholangioscopy (DSOC), one of a newer method of endocanal exploration via ERCP- commonly known as the SpyGlass - helps to provide the visual diagnostics of the strictures based on morphological and vascular patterns and to provide directed intraductal biopsy (SpyBite) from the lesions. The combination of both should increase the diagnostic yield in the evaluation of indeterminate biliary stricture by DSOC.
  ERCP is the most widely used diagnostic procedure in patients with biliary obstruction. It enables to identify the biliary stricture, to determinate its location and help providing tissue sampling from the stricture for cytological evaluation. Different methods were used to take samples from the site of the stenosis. Brushing and endocanal forceps biopsies were the most used techniques. The samples from these two techniques will be additionaly examinated using Fluorescence in Situ Hybridization (FISH).

SUMMARY:
The management of biliary strictures depends on their correct pre-operative evaluation which remains challenging. Despite the emerging multitudes of new diagnostic opportunities and modalities which exist today, there is still a large number of biliary stenosis misdiagnosed with a profound negative impact on the patients´ outcome. The study´s aim is to compare the diagnostic yield of primary peroral cholangioscopy and ERCP (with conventional sampling - brushing and forceps biopsy - completed with the FISH) in patients with suspected malignant stricture of the common bile duct and to evaluate the impact of both methods on the management of patients with biliary stricture.

DETAILED DESCRIPTION:
The management of biliary strictures depends on their correct pre-operative evaluation which remains challenging. Biliary strictures have various etiologies (traumatic, inflammatory, tumoral, ischemic etc), which are necessarily needed to be known for the correct therapeutic approach. Despite the emerging multitudes of new diagnostic opportunities and modalities (laboratory, radiological, endoscopic, histopathologic and immunohistological) which exist today, there is still a large number of biliary stenosis misdiagnosed with a profound negative impact on the patients´ outcome. The dilemma that exists is how to balance the risk of missing the chance of curative surgery for some malignancy and preventing some patients from unnecessary surgery for benign etiologies and not to waste time. Therefore, diagnostic methods which can maximize the chance of the preoperative diagnosis of indeterminate biliary strictures are needed.

This study will:

compare two methods helping in the diagnosis of suspected malignant biliary stricture-SMBS evaluate the impact of both methods on the management of patients with biliary strictures.

* ERCP (Endoscopic retrograde cholangiopancreatography) is the most widely used diagnostic procedure in patients with biliary obstruction. It enables to identify the biliary stricture, to determinate its location and help providing tissue sampling from the stricture for cytological evaluation. Different methods were used to take samples from the site of the stenosis. Brush-cytology and endocanal forceps biopsies were the most used techniques, both with differents specificity a sensitivity. It was demonstrated by different studies, that Fluorescence in Situ Hybridization (FISH) improved the diagnostic yield of routine cytology. That is the reason why the investigators are going to combine FISH with the conventional sampling methods to maximize the chance to determine the etiology of stenosis early and avoid wasting time.
* The peroral cholangioscopy (DSOC), one of a newer method of endocanal exploration via ERCP- commonly known as the SpyGlass - helps to provide the visual diagnostics of the strictures based on morphological and vascular patterns and to provide directed intraductal biopsy (SpyBite) from the lesions. The combination of both methods should increase the diagnostic yield in the evaluation of indeterminate biliary stricture by DSOC. Because of its high costs, the DSOC is mostly provided later, that is when the ERCP cytology failed (secondary DSOC). This wasted time can be important and determinable for the patients´ outcome. So primary cholangioscopy could help in the correct management of patients with indeterminate biliary stricture, without wasting time.

The study will compare the primary DSOC to ERCP. Success (positivity) is defined by the presence of benign or malignant cells, adequate to make the final tissue diagnosis. Another examination should be performed in situations where the initial method failed.

Gold standard for final diagnosis should be the histology from surgery resection. In patients without surgery, clinical evaluation and cross-over methods are used for comparison of initial methods.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected malignant biliary stricture
2. Localization: Extrahepatic biliary duct
3. Patient´s consent with a diagnostic procedure
4. Age : 18 years or more

Exclusion Criteria:

1. Intrahepatic biliary strictures
2. Duodenal stenosis (endoscopically)
3. Age : < 18 years
4. Coagulopathy :

   (INR >1,5, Platelets < 100)
5. Pregnancy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
compare the diagnostic yield of the primary peroral cholangioscopy and the ERCP in patients with suspected malignant biliary stricture - SMBS | 1-7 days
  The the sensitivity (%) and specificity (%) of primary Peroral Cholangioscopy and ERCP(with conventional tissue sampling completed with FISH) in patients with suspected malignant stricture of the common bile duct are evaluated. Success (positivity) is defined by the presence of benign or malignant cells, adequate to make the final tissue diagnosis. Based on the previous studies and the experiences of our endoscopists and pathologist, we can expect the diagnostic yield of primary SpyGlass around 92% and of the second method around 75% in the study population (the samples size 66).
evaluate the impact of both methods on management of patients with biliary stricture. | 3-6 months
  The proportion of patients (%) who will miss the chance of curative surgery for some malignancy and the proportion of patients (%) who will not have unnecessary surgery for benign etiologies are evaluated in each group.
evaluate the cost-effectiveness of both methods on management of patients with biliary stricture. | 3-6 months
  The ratio cost (USD)/diagnostic yield(%) of both methods is evaluated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Urban, MD,pHD, Study Chair — 2nd Department of Internal Medicine, University Hospital Olomouc, Czech Republic
Locations (1):
- 2nd Department of Internal Medicine, University Hospital and Palacký University, Olomouc, Czech Republic, Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No